CLINICAL TRIAL: NCT06397066
Title: Comparative Study of White Light Endoscopy and Magnifying Endoscopy in Assessing the Status of Helicobacter Pylori Infection
Brief Title: White Light Endoscopy and Magnifying Endoscopy in Assessing the Status of Hp Infection
Status: Recruiting | Type: Observational
Sponsor: Jilin University (Other)
Responsible Party: Principal Investigator, Dong Yang, Assisted Investigator, Jilin University
Other Study IDs: 130028
Record Dates: First submitted 2024-04-30; First posted 2024-05-02 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Helicobacter Pylori Infection
Keywords: Hp infection status; magnifying endoscopy; white light endoscopy; immunohistochemical test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the white light endoscopy group: The characteristics of white light endoscopic extraction include degree of atrophy (Kimura-Takemoto classification), congestion and edema, yellow white nodules, mucus turbidity, the arrangement of the collecting veins is regular (RAC)/irregular/disappearing, goose flesh, map-like redness, blood scabs, gastric fundus gland polyps, and scratch syndrome, and are judged according to the Kyoto Classification of Gastritis.
  Interventions: Procedure: White light endoscopy group
- the Magnifying endoscopy group: Magnifying endoscopy(ME) uses Narrow Band Imaging (NBI)+ME to observe the non atrophic area of the gastric fundus gland. According to the proportion of the opening of the gastric fundus gland duct in one magnified field of view, it is classified as grade 1 ≤ 25%, indicating Hp current infection, 25%<grade 2<50%, Hp uncertain state, indicating Hp current infection or after recent sterilization, grade 3 ≥ 50%, indicating Hp non-infection or past H. pylori infection.
  Interventions: Procedure: Magnifying endoscopy group

INTERVENTIONS:
Procedure: White light endoscopy group — White light endoscopy observe the characteristics of mucosa under white light
  Groups: the white light endoscopy group
Procedure: Magnifying endoscopy group — NBI+ME to observe the non atrophic area of the gastric fundus gland. The results depend on the ratio of gastric fundus gland.
  Groups: the Magnifying endoscopy group

SUMMARY:
By comparing the characteristics of Helicobacter pylori (Hp) infection under magnifying endoscopy and white light endoscopy, and making judgments of Hp infection status, the advantages and disadvantages of the two endoscopic examination methods are summarized to improve the accuracy of subsequent endoscopic Hp infection status judgments.

DETAILED DESCRIPTION:
This study adopts a cross-sectional study. The expected recruitment time for all participants is 12 months. Our endoscopy center conducts magnifying staining endoscopy examination, along with endoscopic Hp immunohistochemical testing, and cases that have recently completed carbon-13 or carbon-14 breath tests.

1.Retrospectively enrolled cases from August 1, 2022 to April 30, 2024, who underwent magnifying endoscopic examination with endoscopic Hp immunohistochemical testing result at the Endoscopy Center of the First Hospital of Jilin University. All enrolled cases had carbon-13 or carbon-14 breath tests, excluding cases of total gastric atrophy and endoscopic type A gastritis. The criteria for determining the status of Hp infection: A positive immunohistochemical or 13/carbon-14 breath test result indicates a current Hp infection. If both of immunohistochemical or 13/carbon-14 breath test result are negative, combined with the treatment history for Hp infection and endoscopic manifestations, they are further classified as non-infection or past H. pylori infection. If there is a treatment history for Hp infection or obvious atrophy under the endoscopy in which atrophy degree greater than or equal to Kimura-Takemoto classification C2 ( atrophy exceeding the gastric angle), it is considered as past H. pylori infection. If there is no such manifestation, it is considered Hp non-infection. Extract the relevant characteristics of Hp infection under white light and magnifying endoscopy from continuous inclusion of cases, and determine the Hp infection status separately. The characteristics of white light endoscopic extraction include degree of atrophy (Kimura-Takemoto classification), congestion and edema, yellow white nodules, mucus turbidity, the arrangement of the collecting veins is regular (RAC)/irregular/disappearing, goose flesh, map-like redness, blood scabs, gastric fundus gland polyps, and scratch syndrome, and are judged according to the Kyoto Classification of Gastritis. Magnifying endoscopy uses NBI+ME to observe the non atrophic area of the gastric fundus gland. According to the proportion of the opening of the gastric fundus gland duct in one magnified field of view, it is classified as grade 1 ≤ 25%, indicating Hp current infection, 25%<grade 2<50%, Hp uncertain state, indicating Hp current infection or after recent sterilization, grade 3 ≥ 50%, indicating Hp non-infection or past H. pylori infection. The investigators conduct a comparative study between white light endoscopy and magnifying endoscopy, and conduct subgroup analysis based on Hp infection status.

Based on the characteristics of white light endoscopy and magnifying endoscopy, summarize and sort out the integrated endoscopic Hp infection status judgment process (named the integrated endoscopic judgment).

Prospective enrollment: From May 1, 2024 to December 31, 2024, patients who underwent magnifying endoscopic examination with endoscopic Hp immunohistochemical testing result at the Endoscopy Center of the First Hospital of Jilin University. All enrolled cases had carbon-13 or carbon-14 breath tests, excluding cases of total gastric atrophy and endoscopic type A gastritis. Using the white light endoscopy, magnifying endoscopy, and integrated endoscopic judgment to determine the Hp infection status, three different endoscopic Hp judgment results will be obtained, and data comparison conducted between the three groups.

All enrolled cases were evaluated blindly by two doctors. If there was no consensus, the third doctor would further evaluate and determine the Hp infection status under white light endoscopy, magnifying endoscopy, and integrated endoscopic judgment. Based on the comparison results, a more accurate endoscopic method will be selected to determine the Hp infection status.

ELIGIBILITY:
Inclusion Criteria:

- Our endoscopy center conducts magnifying staining endoscopy examination, along with endoscopic Hp immunohistochemical testing, and cases that have recently completed carbon-13 or carbon-14 breath tests.

Exclusion Criteria:

- Total gastric atrophy and endoscopic type A gastritis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Our endoscopy center conducts magnifying staining endoscopy examination, along with endoscopic Hp immunohistochemical testing, and cases that have recently completed carbon-13 or carbon-14 breath tests.
Sampling Method: Probability Sample
Enrollment: 168 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of different observation method | at the end of the observation of endoscopy procedure
  white light endoscopy, magnifying endoscopy, and integrated endoscopic judgment to determine the status of Hp infection (including Hp current infection, Hp negative, and past H. pylori infection status)

SECONDARY OUTCOMES:
Sensitivity of different observation method | at the end of the observation of endoscopy procedure
  white light endoscopy, magnifying endoscopy, and integrated endoscopic judgment to determine the status of Hp infection (including Hp current infection, Hp negative, and past H. pylori infection)
specificity of different observation method | at the end of the observation of endoscopy procedure
  white light endoscopy, magnifying endoscopy, and integrated endoscopic judgment to determine the status of Hp infection (including Hp current infection, Hp negative, and past H. pylori infection)
result of immunohistochemistry | the end of enrollment
  Biopsy of Helicobacter pylori from the large and small curvature of the gastric antrum and the large and small curvature of the gastric body, and submission for immunohistochemical detection
result of breath tests. | the end of enrollment
  the results of carbon-13 or carbon-14 breath tests showed the Hp infection status

CONTACTS AND LOCATIONS:
Overall Officials: Dong Yang, doctor, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- the First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No